CLINICAL TRIAL: NCT05471323
Title: A Single-arm, Single/Multiple Dose-escalation and Dose-extension Phase I Clinical Trial of RC1012 Injection (Allogeneic DNT Cells) in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Phase I Clinical Trial of RC1012 Injection in Patients With r/r AML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Ruishun Biotech Co., Ltd (Industry)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC1012-AML001
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: r/r AML; Cell Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC1012 injection (allo-DNT Cells) (Experimental): Experimental: RC1012 injection (allo-DNT Cells) The trial is divided into two parts: Part A1 is a single- dose escalation trial with three dose groups (5×10^7 cells/kg, 1.5×10^8 cells/kg, 4.5×10^8 cells/kg), with 9-18 patients planned to be enrolled. Part A2 is a multiple-dose escalation trial consisting of 2 dose groups (1.5×10^8 cells/kg and 4.5×10^8 cells/ kg at day 0, day 7 and day 14), with 9-12 patients planned to be enrolled. Part B is a multiple-dose extension trial in which the Safety Review Committee evaluates whether to extend an additional 3-6 patients to receive the multiple cell infusions based on available PK and safety data.
  Interventions: Biological: RC1012 injection (allo-DNT cells)

INTERVENTIONS:
Biological: RC1012 injection (allo-DNT cells) — RC1012 injection (allo-DNT cells) from healthy donors and have been proved to be safe and demonstrated potent cytotoxicity against AML blasts from AML patients in preclinical and preliminary clinical studies. Allo- DNT cells will be collected from healthy donors (NO MHC match needed) and injected into patients. The drug for this study is an off-the-shelf product. Patients DO NOT need to wait for the cell manufacturing.

SUMMARY:
To evaluate the safety and tolerability of RC1012 infusion in patients with relapsed or refractory Acute Myelocytic Leukemia (r/r AML).

DETAILED DESCRIPTION:
This study aims to evaluate the safety and tolerability of RC1012 injection in patients with relapsed or refractory Acute Myelocytic Leukemia (r/r AML).

DNT cells are mature T lymphocytes that comprise 3-10% of T cells in human peripheral blood mononuclear cells (PBMC). Allo-DNT cells from healthy donors have been proved to be safe and demonstrated potent cytotoxicity against AML blasts from AML patients in preclinical and preliminary clinical studies. Allo-DNT cells will be collected from healthy donors (NO MHC match needed) and infused into patients. The drug for this study is an off-the-shelf product. Patients DO NOT need to wait for the cell manufacturing.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an ICF and expect to complete the study procedures for follow-up examinations and treatment.
2. Aged 18 to 70 years (including cut-offs), regardless of gender.
3. Accordance with the diagnostic criteria of AML in the 2016 WHO staging and meeting the diagnostic criteria of relapsed and refractory in the Chinese Guidelines for the Treatment of Relapsed/Refractory Acute Myeloid Leukemia (2017 edition).

   * Diagnostic criteria for Relapsed AML: reappearance of leukemic cells in peripheral blood or >5% primitive/naive cells in bone marrow after CR (except for other causes such as bone marrow regeneration after consolidation chemotherapy) or extra-marrow infiltration of leukemic cells.
   * Diagnostic criteria for refractory AML: primary refractory disease that has not achieved complete remission after two courses of induction chemotherapy with a standard regimen (containing cytarabine and an anthracycline or anthraquinone).
4. The patient has recovered from the toxicity of the prior treatment, i.e., less than a grade 2 CTCAE toxicity rating (unless the abnormality is tumor-related).
5. ECOG score 0 to 1.
6. Appropriate organ function, and accordance with the following criteria within 7 days prior to lymphodepleting chemotherapy.

   * Glutathione aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN)
   * Glutamic aminotransferase (ALT) ≤ 3 times ULN.
   * Total bilirubin ≤ 1.5 times ULN, unless the patient has documented Gilbert syndrome. Patients with Gilbert-Meulengracht syndrome with total bilirubin ≤ 3.0 times ULN and direct bilirubin ≤ 1.5 times ULN may be included.
   * Serum creatinine ≤ 1.5 times ULN or a creatinine clearance ≥ 60 ml/min.
   * Hemoglobin ≥ 60 g/L or hemoglobin maintained at that level following transfusion.
   * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L.
   * A platelet count ≥ 30 x 10^9/L or a platelet count maintained at that level following a platelet transfusion
   * Left ventricular ejection fraction (LVEF) ≥ 45%.
7. Female patients with of childbearing potential should have a negative pregnancy test during the screening period. Any male and female patients of childbearing potential must agree to use an effective contraception method for at least six months from the time that they sign the informed consent form until the end of the cell infusion. Female patients without childbearing potential (meeting at least 1 of the following criteria) is described below.

   * Have undergone a hysterectomy or bilateral oophorectomy
   * Medically recognized as ovarian failure.
   * Medically recognized as post-menopausal (at least 12 consecutive months of menopause without pathological or physiological cause).

Exclusion Criteria:

1. A diagnosis of acute promyelocytic leukemia.
2. Patients with extramedullary infiltration of leukemia.
3. Evidence or history of central nervous system invasion or cranial neuropathy.
4. Patients with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titration assay not within the normal reference range, positive hepatitis C virus (HCV) antibody and peripheral blood HCV RNA ,positive for human immunodeficiency virus (HIV), or positive for cytomegalovirus (CMV) DNA, or positive syphilis test.
5. Persons with hypersensitivity to excipients of RC1012 injection (e.g., human albumin) or other drugs recommended in the study protocol (e.g., lymphodepleting treatment, Tocilizumab).
6. Serious cardiac disease, including but not limited to severe arrhythmia, unstable angina, massive heart attack, New York Heart Association class III or IV cardiac insufficiency, refractory hypertension.
7. Persons who have previously received an organ transplant or are preparing to receive an organ transplant (except for hematopoietic stem cell transplantation)
8. Persons with acute and chronic graft-vs-host disease (GVHD)
9. Those who have received a hematopoietic stem cell transplant within 2 months prior to screening tests.
10. Active neurological autoimmune or inflammatory diseases (e.g. Guillain-Barre Syndrome (GBS), Amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular disease (e.g. cerebral oedema, Posterior Reversible Encephalopathy Syndrome (PRES)).
11. Patients with a life expectancy of less than 3 months
12. Patients have been involved in other clinical studies within 3 months prior to screening.
13. Patients, in the judgement of the investigator and/or clinical criteria, are contraindicated to any study procedure or have other medical conditions that may place them at unacceptable risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of allo-DNT Cell Therapy for Relapsed/Refractory Acute Myelocytic Leukemia
Maximum Tolerated Dose (MTD) | Up to 28 days
  MTD was the highest dose for DLT in ≤1/6 subjects
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) indicator (Cmax) | Up to 90 days
  The peak concentration of allo-DNT cells amplified in the peripheral blood (Cmax, detected by Flow Cytometry).
Pharmacokinetics (PK) indicator (AUC) | Up to 2 years
  Allo-DNT cells blood concentrations will be measured at different time points to evaluate the area under the curve (AUC). (AUC, detected by Flow Cytometry).
Pharmacokinetics (PK) indicator (Tmax) | Up to 2 years
  Allo-DNT cells blood concentrations will be measured at different time points to evaluate the peak time (Tmax) in peripheral blood. Tmax is defined as the time to reach the highest concentration (Tmax, detected by Flow Cytometry).
Pharmacokinetics (PK) indicator (T1/2) | Up to 2 years
  Allo-DNT cells blood concentrations will be measured at different time points to evaluate the elimination half-life in hours (T1/2). T1/2 is defined as the time point when the concentration of allo-DNT reaches half of maximum in a patient's peripheral blood (T1/2, detected by Flow Cytometry).
Overall Response Rate | Up to 2 years
  ORR includes complete response (CR), CRi and PR. CR was defined as < 5% bone marrow blasts in an aspirate with spicules, no blasts with Auer rods or persistence of extramedullary disease, and independent of transfusions; CRi: was defined as<5% bone marrow blasts, either ANC<1×10^9/L or platelets<100×10^9/L, transfusion independence but with persistence of cytopenia; PR was defined as decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow aspirate and the normalization of blood counts.
Event-Free Survival | Up to 2 years
  From the date of enrollment in the clinical trial until the failure of treatment, relapse or death.
Duration of Response | Up to 2 years
  The time from the start of the first assessment of CR or PR to the first assessment as disease recurrence or progression or death
Relapse-Free Survival | Up to 2 years
  Relapse-free survival is the time from study enrollment until documented disease relapse, or death from any cause.
Overall Survival | Up to 5 years
  From the date of entry into the clinical study until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Cai, MD, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China